CLINICAL TRIAL: NCT02439515
Title: Fall Prevention and Locomotion Recovery in Post-stroke Patients: A Multimodal Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Salvatore Maugeri (Other)
Collaborators: Politecnico di Milano (Other)
Responsible Party: Principal Investigator, Simona Ferrante, PhD, Politecnico di Milano
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GR-2010-2312228-SF
Record Dates: First submitted 2015-04-24; First posted 2015-05-08 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Stroke
Keywords: post-acute stroke; functional electrical stimulation; biofeedback; balance; cycling; rehabilitation; gait
MeSH Terms: conditions — Stroke | interventions — Recruitment Detection, Audiologic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Biofeedback training (Experimental): It consists of 15 daily sessions of voluntary cycling training augmented by functional electrical stimulation (FES) followed by 15 daily sessions of balance training (multimodal biofeedback training). Both cycling and balance training are supported by a visual biofeedback and last about 20 minutes.
  In addition to cycling or balance training, subjects perform standard physical therapy in order to reach 90 minutes of training per day.
  Interventions: Device: Cycling; Device: Balance; Other: Standard physical therapy
- Usual Care (Active Comparator): It consists of 30 daily sessions of standard physical therapy. Each session last about 90 minutes.
  Interventions: Other: Standard physical therapy

INTERVENTIONS:
Device: Cycling — Voluntary cycling augmented by electrical stimulation and biofeedback
  Other Names: MOTOmed, Reck GmbH; PowerForce system, Radlabor GmbH; RehaStim; Hasomed GmbH
  Arms: Biofeedback training
Device: Balance — Balance control exercises with visual biofeedback
  Other Names: Balance board basic™, NeuroCom® International, Inc.
  Arms: Biofeedback training
Other: Standard physical therapy — It consists of stretching, muscular conditioning, exercises for trunk control, standing, and walking training, and upper limb rehabilitation.

SUMMARY:
The study proposes a novel rehabilitative program for the recovery of locomotor abilities in post-acute stroke patients. The hypothesis is that a rehabilitative program which involves a biofeedback cycling training combining voluntary effort and Functional Electrical Stimulation (FES) of the leg muscles, and a biofeedback balance training is superior to usual care in improving walking abilities, disability, motor performance, and independence of post-acute stroke patients. The innovative approach is to investigate whether interventions which do not directly involve locomotor functions but movements similar in terms of kinematic patterns and neural commands (e.g. pedaling), or aimed at recovering an essential prerequisite for walking, such as postural control during upright stance, may improve and/or accelerate the recovery of walking abilities.

A single-blind randomized controlled study is carried out. Participants are post-acute stroke patients experiencing a first stroke less than 6 months before recruitment, with an adult age, a low level of spasticity of the leg muscles (Modified Ashworth scale <2), no limitations at hip, knee, and ankle joints, and able to sit up to 30 minutes. Subjects are randomized to one of two groups, one performing the novel rehabilitative program in addition to usual care (experimental group), and one performing usual care alone (control group).

The experimental program consists of 15 sessions of FES-supported voluntary cycling training followed by 15 sessions of balance training. Both cycling and balance training are supported by a visual biofeedback in order to maximize patients' involvement in the exercise and are performed in addition to usual care.

The control group is involved in standard physical therapy which includes stretching, muscular conditioning, exercises for trunk control, standing, and walking training, and upper limb rehabilitation.

Both training programs last 6 weeks and patients are trained daily for about 90 minutes. Cycling and balance training last about 20 minutes; thus, patients in the experimental group perform only about 70 minutes of usual care.

Participants are evaluated at baseline (T1), after the end of the cycling training or after 3 weeks of usual care (post-treatment, T2), after the end of the whole intervention (post-treatment, T3), and about 6 months after the end of the intervention (follow-up, T4).

DETAILED DESCRIPTION:
More details on the experimental training program are here provided.

The cycling training is performed on a motorized cycle-ergometer (MOTOmed, Reck GmbH) equipped with force sensors mounted at the base of the cranks (PowerForce system, Radlabor GmbH). The acquired force signals are displayed to the subjects who are asked to achieve a symmetrical involvement of the two legs. To deliver FES, a current-controlled 8-channel stimulator (RehaStim; Hasomed GmbH) is used and surface electrodes are applied in a bipolar configuration on the quadriceps, hamstrings, gastrocnemius lateralis, and tibialis anterior of both legs. Rectangular biphasic pulses with a pulse width of 400 μs and a stimulation frequency of 20 Hz are adopted. The stimulus intensity is set on each muscle the first day of training: for the paretic muscles values well tolerated by the subject and able to produce visibly good muscle contractions are identified, whereas for the healthy side lower values just above the sensory threshold are used. The stimulation timing is synchronized to the cycling movement according to physiological stereotyped activation patterns.

The balance training is performed during upright stance using a balance board (Balance board basic™, NeuroCom® International, Inc.). Subjects are asked to keep still or move their center of pressure following a target displayed on a screen in front of them.

ELIGIBILITY:
Inclusion Criteria:

* post-acute stroke patients experiencing a first stroke (both ischemic or hemorrhagic) less than 6 months before recruitment
* low level of spasticity of the leg muscles (Modified Ashworth scale <2)
* no limitations at hip, knee, and ankle joints
* able to sit up to 30 minutes

Exclusion Criteria:

* neurological impairment (Mini mental scale <24)
* presence of other neurological diseases
* spatial hemineglect
* cardiac pacemakers
* allergy to electrodes
* an inability to tolerate electrical stimulation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-07 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Gait Speed | "6 weeks"
  Subjects are asked to walk three times at self-selected speed over the GaitRite mat using their walking aid (if any) or receiving the needed assistance. Spatial-temporal parameters are evaluated using the GaitRite software.

SECONDARY OUTCOMES:
Gait speed | "Day 0", "3 weeks", "6 months+6 weeks"
  Subjects are asked to walk three times at self-selected speed over the GaitRite mat using their walking aid (if any) or receiving the needed assistance. Spatial-temporal parameters are evaluated using the GaitRite software.
Aerobic capacity/endurance during gait assessed by 6-minute walking test | "Day 0", "3 weeks", "6 weeks", "6 months+6 weeks"
  Subjects are asked to walk along a rectilinear corridor for 6 minutes. The distance covered is measured.
Motor power of the paretic lower extremity assessed by Motricity Index | "Day 0", "3 weeks", "6 weeks", "6 months+6 weeks"
  Italian version; Only leg-subscale of the paretic side
Trunk Control assessed by Trunk Control Test | "Day 0", "3 weeks", "6 weeks", "6 months+6 weeks"
  Italian version
Abilities during activities of daily life assessed by Functional Independence Measure | "Day 0", "3 weeks", "6 weeks", "6 months+6 weeks"
  Italian version
Risk of fall assessed by Fall Efficacy Scale | "Day 0", "3 weeks", "6 weeks", "6 months+6 weeks"
  Italian version
Balance control assessed by Berg Balance Scale | "Day 0", "3 weeks", "6 weeks", "6 months+6 weeks"
  Italian version
Patient's perception of the effect of the intervention assessed by Global Perceived Effect | "6 weeks"
  Italian version
Pedaling performance assessed by Pedaling test | "Day 0", "3 weeks","6 months+6 weeks"
  A pedaling test is performed on the motorized cycle-ergometer to measure the force produced by the two sides during voluntary cycling as well as electromyography activations of the main lower limb muscles. Subjects are asked to pedal at four difference target pace (20 RPM, 30 RPM, 40 RPM, and 50 RPM), while the ergometer motor maintains a constant cadence of 10 RPM less than the target. A visual numerical cadence indicator and a metronome help the subjects to keep the constant cadence.
Balance performance assessed by Balance test | "3 weeks", "6 weeks", "6 months+6 weeks"
  Postural stability is evaluated using the commercial balance board exploited in the experimental intervention program (Balance board basic™, NeuroCom® International, Inc.). Pre-defined assessments are used to evaluate the postural sways during upright stance both with eyes open and closed; the limits of stability in all directions (forward, backward, right, and left); and the capability to shift the weight both left/right and forward/backward.

CONTACTS AND LOCATIONS:
Overall Officials: Simona Ferrante, PhD, Principal Investigator — Politecnico di Milano
Locations (1):
- Istituti Clinici e Scientifici Maugeri, Lissone, Monza Brianza, Italy

REFERENCES:
- [Background] Ambrosini E, Ferrante S, Ferrigno G, Molteni F, Pedrocchi A. Cycling induced by electrical stimulation improves muscle activation and symmetry during pedaling in hemiparetic patients. IEEE Trans Neural Syst Rehabil Eng. 2012 May;20(3):320-30. doi: 10.1109/TNSRE.2012.2191574. Epub 2012 Apr 13. PMID 22514205
- [Background] Ferrante S, Ambrosini E, Ravelli P, Guanziroli E, Molteni F, Ferrigno G, Pedrocchi A. A biofeedback cycling training to improve locomotion: a case series study based on gait pattern classification of 153 chronic stroke patients. J Neuroeng Rehabil. 2011 Aug 24;8:47. doi: 10.1186/1743-0003-8-47. PMID 21861930
- [Background] Ambrosini E, Ferrante S, Pedrocchi A, Ferrigno G, Molteni F. Cycling induced by electrical stimulation improves motor recovery in postacute hemiparetic patients: a randomized controlled trial. Stroke. 2011 Apr;42(4):1068-73. doi: 10.1161/STROKEAHA.110.599068. Epub 2011 Mar 3. PMID 21372309
- [Derived] Ambrosini E, Parati M, Peri E, De Marchis C, Nava C, Pedrocchi A, Ferriero G, Ferrante S. Changes in leg cycling muscle synergies after training augmented by functional electrical stimulation in subacute stroke survivors: a pilot study. J Neuroeng Rehabil. 2020 Feb 27;17(1):35. doi: 10.1186/s12984-020-00662-w. PMID 32106874
- [Derived] Ambrosini E, Peri E, Nava C, Longoni L, Monticone M, Pedrocchi A, Ferriero G, Ferrante S. A multimodal training with visual biofeedback in subacute stroke survivors: a randomized controlled trial. Eur J Phys Rehabil Med. 2020 Feb;56(1):24-33. doi: 10.23736/S1973-9087.19.05847-7. Epub 2019 Sep 26. PMID 31556542